CLINICAL TRIAL: NCT04267406
Title: Investigation of Changes in ADAMTS-13 and Von Willebrand Factor Levels and Activities in Children With Cirrhosis and/or Portal Hypertension
Brief Title: ADAMTS-13 and Von Willebrand Factor Levels and Activities in Children With Cirrhosis and/or Portal Hypertension
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ali Islek, Associate Professor, Ataturk University
Other Study IDs: 218S871
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Coagulation Disorder; Cirrhosis, Liver
Keywords: Von willebrand factor; ADAMTS-13; Children; Cirrhosis; Portal hypertension
MeSH Terms: conditions — Hemostatic Disorders; Liver Cirrhosis; Fibrosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cirrhosis: Patients who diagnosed as cirrhosis. 2 ml EDTA blood sample was taken from patients during their routine controls or at the time of diagnosis. Samples will be tested for ADAMTS-13 and vWF levels and activity at the end of study.
- Non-cirrhotic portal hypertension: Patients who diagnosed as extrahepatic portal hypertension (due to portal vein thrombosis). 2 ml EDTA blood sample was taken from patients during their routine controls or at the time of diagnosis. Samples will be tested for ADAMTS-13 and vWF levels and activity at the end of study.
- Control: Healthy volunteers, who admitted to our hospital for any complaints, but was not determined any organic disease. 2 ml EDTA blood sample was taken from healthy volunteers, during their hospital admition. Samples will be tested for ADAMTS-13 and vWF levels and activity at the end of study.

SUMMARY:
Hemostasis-related disorders are common in cirrhosis and portal hypertension. However, it is not known whether the net effect of changes in hemostasis in the sense of predisposition to hemorrhagic or thrombotic state. It is suggested that increasing the concentration and activities of Von Willebrand factor (vWF) and decline ADAMTS-13 (A Disintegrin and Metalloproteinase with Trombospondin type 1 motif, member 13) may cause thrombophilic changes in cirrhosis and portal hypertension. The aim of this study was to investigate the changes in ADAMTS-13 (A disintegrin and metalloproteinase with thrombospondin motifs 13) and von willebrand factor (vWF) levels and activities in patients with cirrhosis and portal hypertension.

DETAILED DESCRIPTION:
Patients of 3 months to 18 years of age, followed-up or newly diagnosed in pediatric gastroenterology unit, who had cirrhosis or non cirrhotic portal hypertension included to the study. Written informed consent obtained from the parents and/or patients. The subjects was grouped in three. The first group consisted of patients with cirrhosis (with or without portal hypertension). The second group consisted of patients with non-cirrhotic portal hypertension (developed due thrombosis of portal vein). The last group consisted of healthy volunteers.

2 ml of EDTA blood was taken from the patients and healty volunters. Samples will be tested for vWF and ADAMTS-13 levels and activities at the end of the study.

The clinical scoring methods, PELD, MELD and Child Pugh scores, treatments received by patients, data from endoscopic, radiological screening, and blood analysis of patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

• Patients with cirrhosis or portal hypertension aged 3 months to 18 years.

Exclusion Criteria:

* Being treated with fresh frozen plasma in the recent month.
* Patients previously diagnosed with bleeding diathesis.
* The patients who consumed vitamin K in the recent three weeks.
* Patients previously diagnosed with another chronic disease (such as renal failure, heart failure etc).
* Patients who suffer from acute or chronic infectious diseases.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with cirrhosis and/or portal hypertension who were treated in Pediatric Gastroenterology Department of Ataturk University Hospital included to the study.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Measuring ADAMTS-13 enzyme levels in collected EDTA bloods. | First day
  Measuring ADAMTS-13 antigen levels using commercial ELISA kits (IU/mL) in all groups.
Measuring ADAMTS-13 activities in collected EDTA bloods. | First day
  Measuring ADAMTS-13 activities using commercial ELISA kits (as a percentage) in all groups.
Measuring vWF antigen levels in collected EDTA bloods. | First day
  Measuring vWF antigen levels using immunoturbidimetric assay (as a percentage) in all groups.
Measuring vWF activities in collected EDTA bloods. | First day
  Measuring vWF activities [von Willebrand factor ristocetin cofactor (vWF:RCo)] by the aggregation of platelets in the presence of ristocetin using immunoturbidimetric assay (as a percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Islek, MD, Principal Investigator — Ataturk University School of Medicine
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lisman T, Caldwell SH, Burroughs AK, Northup PG, Senzolo M, Stravitz RT, Tripodi A, Trotter JF, Valla DC, Porte RJ; Coagulation in Liver Disease Study Group. Hemostasis and thrombosis in patients with liver disease: the ups and downs. J Hepatol. 2010 Aug;53(2):362-71. doi: 10.1016/j.jhep.2010.01.042. Epub 2010 May 12. PMID 20546962
- [Background] Plaimauer B, Zimmermann K, Volkel D, Antoine G, Kerschbaumer R, Jenab P, Furlan M, Gerritsen H, Lammle B, Schwarz HP, Scheiflinger F. Cloning, expression, and functional characterization of the von Willebrand factor-cleaving protease (ADAMTS13). Blood. 2002 Nov 15;100(10):3626-32. doi: 10.1182/blood-2002-05-1397. Epub 2002 Jul 12. PMID 12393399
- [Background] Turner NA, Nolasco L, Ruggeri ZM, Moake JL. Endothelial cell ADAMTS-13 and VWF: production, release, and VWF string cleavage. Blood. 2009 Dec 3;114(24):5102-11. doi: 10.1182/blood-2009-07-231597. Epub 2009 Oct 12. PMID 19822897
- [Result] Goel A, Alagammai PL, Nair SC, Mackie I, Ramakrishna B, Muliyil J, Keshava SN, Eapen CE, Elias E. ADAMTS13 deficiency, despite well-compensated liver functions in patients with noncirrhotic portal hypertension. Indian J Gastroenterol. 2014 Jul;33(4):355-63. doi: 10.1007/s12664-014-0460-4. Epub 2014 Apr 24. PMID 24756423
- [Result] Uemura M, Fujimura Y, Matsumoto M, Ishizashi H, Kato S, Matsuyama T, Isonishi A, Ishikawa M, Yagita M, Morioka C, Yoshiji H, Tsujimoto T, Kurumatani N, Fukui H. Comprehensive analysis of ADAMTS13 in patients with liver cirrhosis. Thromb Haemost. 2008 Jun;99(6):1019-29. doi: 10.1160/TH08-01-0006. PMID 18521503
- [Result] Lisman T, Bongers TN, Adelmeijer J, Janssen HL, de Maat MP, de Groot PG, Leebeek FW. Elevated levels of von Willebrand Factor in cirrhosis support platelet adhesion despite reduced functional capacity. Hepatology. 2006 Jul;44(1):53-61. doi: 10.1002/hep.21231. PMID 16799972